CLINICAL TRIAL: NCT02681978
Title: Heart Rate Reduction by IVabradine for Improvement of ENDothELial Function in Patients With Coronary Artery Disease: the RIVENDEL Study
Brief Title: Ivabradine to Improve Endothelial Function in Patients With Coronary Artery Disease
Acronym: RIVENDEL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Germano Di Sciascio, Prof. Germano Di Sciascio, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RIVENDEL
Record Dates: First submitted 2016-02-04; First posted 2016-02-15 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ivabradine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ivabradine group (Active Comparator): Ivabradine 5 mg twice daily + standard medical therapy
  Interventions: Drug: Ivabradine; Drug: Standard medical therapy
- Control group (Other): Standard medical therapy
  Interventions: Drug: Standard medical therapy

INTERVENTIONS:
Drug: Ivabradine — Ivabradine 5 mg twice daily
  Arms: Ivabradine group
Drug: Standard medical therapy — Standard medical therapy for patients with coronary artery disease undergoing percutaneous coronary interventions

SUMMARY:
This study evaluates the effect of ivabradine on endothelial function in patients with coronary artery disease (CAD) after complete revascularization with percutaneous coronary angioplasty (PCI). At least 30 days after PCI, patients will be randomized to receive ivabradine 5 mg twice daily or to continue with standard medical therapy.

ELIGIBILITY:
Inclusion Criteria:

* history of stable coronary disease
* complete coronary revascularization with PCI at least 1 month prior to recruitment
* sinus rhythm
* absence of anginal symptoms

Exclusion Criteria:

* resting heart rate <60 beats per minute
* severe reduction of left ventricle ejection fraction (<40%)
* coronary artery by-pass surgery
* myocardial infarction, stroke or cerebral transient ischemic attack within the previous 6 months
* implanted pacemaker, cardioverter, or defibrillator
* sick sinus syndrome
* sinoatrial block
* congenital long QT
* complete atrioventricular block

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Flow-mediated dilation of the brachial artery | 8 weeks

SECONDARY OUTCOMES:
Number of patients with flow-mediated dilation of the brachial artery <7% | 8 weeks
Endothelium-independent dilation of the brachial artery | 8 weeks
  Dilation of the brachial artery after administration of 0.5 mg sublingual nitroglycerin
Correlation between heart rate and flow-mediated dilation of the brachial artery | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Mangiacapra, MD, PhD, Principal Investigator — Campus Bio-Medico University
Locations (1):
- Campus Bio-Medico University, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mangiacapra F, Colaiori I, Ricottini E, Balducci F, Creta A, Demartini C, Minotti G, Di Sciascio G. Heart Rate reduction by IVabradine for improvement of ENDothELial function in patients with coronary artery disease: the RIVENDEL study. Clin Res Cardiol. 2017 Jan;106(1):69-75. doi: 10.1007/s00392-016-1024-7. Epub 2016 Aug 12. PMID 27520989